CLINICAL TRIAL: NCT06385353
Title: Baseline Ultrasound Venous Thrombosis Burden and the Risk of Post-thrombotic Syndrome in Patients With a First Acute Episode of Symptomatic Deep Vein Thrombosis of the Lower Limbs - The "DVT-Burden" Project -
Brief Title: DVT Burden and the Risk of Post-thrombotic Syndrome
Acronym: DVT-Burden
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Assistance Publique Hopitaux De Marseille (Other); F-CRIN INNOVTE Research Network (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-CHITS-003; 2023-A02652-43 (Other: ID-RCB number)
Record Dates: First submitted 2024-04-16; First posted 2024-04-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Postthrombotic Syndrome
Keywords: Venous thrombosis; Thrombus burden; Ultrasonography; Thrombus resolution; Post-thrombotic syndrome
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Association between thrombosis burden and occurrence of PTS (Experimental)
  Interventions: Other: Quantification of deep vein thrombosis burden and assessment of post-thrombotic syndrome

INTERVENTIONS:
Other: Quantification of deep vein thrombosis burden and assessment of post-thrombotic syndrome — Post-thrombotic syndrome will be assessed by the Villalta score until 6 months of follow-up.
  Data collected from colour doppler ultrasound will be used to calculate the Venous Volumetric Index to quantify deep vein thrombosis burden until 6 months of follow-up.

SUMMARY:
Post-thrombotic syndrome (PTS) is the most common chronic complication of deep vein thrombosis (DVT), with major consequences for patient quality of life and cost of management. Identifying patients at high risk of developing PTS could be useful for its prevention and may lead to more appropriate therapeutic strategies to reduce its incidence and severity.

Prognostic tools for predicting risk are very useful for choosing the optimum treatment and improving patient management and are a preliminary step before developing predictive models useful for determining sensitivity to treatment. At present, although several prognostic markers and models have been proposed, it is still difficult to predict who will develop a PTS or a moderate to severe PTS. The development of PTS is multifactorial and depends largely on the extent and severity of venous obstruction which supports the theory of thrombosis burden (DVT-Burden) as a potential prognostic marker for PTS. It therefore seems important to study the association between thrombosis burden and the occurrence of PTS.

The Venous Volumetric Index or VVI (Ouriel 1999) will be used for quantifying DVT-Burden. The VVI was constructed by calculating the volume from the diameter and length of 14 venous segments from the calf veins to the inferior vena cava. The VVI has been validated for its ability to discriminate between symptomatic and asymptomatic DVT and has shown superior performance to other methods for quantifying DVT.

This study aim to assess the performance of baseline DVT-burden estimated by the VVI score on ultrasound for predicting the occurrence and the severity of PTS as assessed by the Villalta scale at 6 months.

DETAILED DESCRIPTION:
This is a multicenter prospective cohort study aiming at assessing baseline DVT-Burden and other prognostic factors for predicting the occurrence and the severity of PTS.

Patients diagnosed with a first episode of DVT of the lower limbs are recruited in offices and departments of vascular medicine. They will be informed of the study by their physician. If patients agree to take part and meet the eligibility criteria, they will be included consecutively in the study after signing an informed consent form.

The study will include follow-up visits at one week (D7±2, for patients participating in the biological research only), 1 month (D30±5), 3 months (D90±5) and 6 months (D180±5).

At each visit, the following examinations will be carried out:

* Assessment of symptoms and clinical signs to evaluate the Villalta score.
* Venous ultrasound evaluation of the lower limbs by colour Doppler ultrasound (CDUS). Data collected will be useful to calculate the VVI score planned at the study analysis phase.

At the D0, D7, D30 and D90 visits, blood samples will be taken for research purposes to assess factors of inflammation, coagulation and fibrinolysis.

At the D90 and D180 visits, the patient will also be asked to complete the VEINES-QOL and SF-36 quality of life questionnaires.

The patient's participation in the research will end at the end of the D180 visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with symptomatic acute deep venous thrombosis of the lower limbs confirmed by ultrasound on the criteria of venous incompressibility and direct image of the thrombus (patients with stable pulmonary embolism associated with a symptomatic deep venous thrombosis can be included)
3. Affiliates or beneficiaries of a social security scheme.

Exclusion Criteria:

1. Pregnant women, women in labour or breastfeeding mothers.
2. Pulmonary embolism haemodynamically unstable defined by systolic blood pressure < 90 mmHg or a drop in systolic blood pressure of at least 40 mmHg during at least 15 min, shock or cardiac arrest.
3. Asymptomatic venous thrombosis.
4. Symptomatic venous thrombosis of both lower limbs (patients with bilateral deep venous thrombosis but symptomatic on one side only can be included).
5. History of ipsilateral or contralateral venous thrombosis of the lower limb.
6. Fracture or orthopedic surgery of the lower limbs in the last 3 months.
7. Dependance caused by age or secondary to a chronic affection, going from the inability to stand up or walk alone without help to bed or armchair rest over.
8. Prophylactic or therapeutic anticoagulant treatment > 5 days.
9. Expected duration of anticoagulant treatment < 3 months (all patients must have a minimum treatment of 3 months).
10. Patient estimated at high risk of bleeding according to investigator clinical judgment (renal, platelet, digestive, hepatic, neurological... origin) .
11. Indication for interruption of the inferior vena cava or venous recanalisation (endovascular, thrombolysis or surgery).
12. Refusal or inability to give written informed consent to participate in the study.
13. Life expectancy < 6 months.
14. Patients under legal protection (guardianship, curatorship, etc.) or safeguard of justice.
15. Patients taking part in a research project for venous thromboembolism that can interfere with the conduct of DVT-BURDEN research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Presence of moderate to severe Post-thrombotic Syndrome (PTS) | 6 months
  The primary outcome measure is the presence of moderate or severe PTS at 6 months as determined by a Villalta score ≥ 10 or the presence of an ulcer. The Villalta score considers items based on symptoms and clinical signs, including skin complications, each assessed on a scale from 0 to 3. The Villalta score is used to diagnose PTS and categorise its severity, according to international recommendations.
  Thrombosis burden is assessed using the VVI index as well as prognostic factors at baseline.
Thrombosis burden | Baseline
  Thrombosis burden is assessed using the Venous Volumetric Index (VVI) as well as prognostic factors at baseline.

SECONDARY OUTCOMES:
Presence of moderate to severe PTS adjusted to other prognostic factors at baseline | 6 months
  PTS is assessed at 6 months by the Villalta scale.
Thrombosis burden adjusted to other prognostic factors at baseline | Baseline
  Thrombosis burden is assessed using the VVI index as well as prognostic factors at baseline.
Presence of moderate to severe PTS adjusted to other prognostic factors at baseline and during follow-up | Baseline, 1 week, 1 month, 3 months and 6 months
  PTS is assessed at 6 months by the Villalta scale. Other prognostic factors related to anticoagulant therapy and compression are assessed during follow-up.
Thrombosis burden adjusted to other prognostic factors at baseline and during follow-up | Baseline, 1 week, 1 month, 3 months and 6 months
  Thrombosis burden is assessed using the VVI index as well as prognostic factors at baseline.
  Other prognostic factors related to anticoagulant therapy and compression are assessed during follow-up.
Time to complete resolution of the thrombus as a function of thrombosis burden at baseline | up to 6 months
Presence of moderate to severe PTS at baseline and at follow-up visits | Baseline, 1 week, 1 month, 3 months and 6 months
  PTS is assessed by the Villalta scale.
Thrombosis burden at baseline and at follow-up visits | Baseline, 1 week, 1 month, 3 months and 6 months
  The thrombus burden is assessed by the VVI index.

OTHER OUTCOMES:
Disease specific health related quality of life | 3 months and 6 months
  Disease specific health related quality of life will be assessed by the Venous Insufficiency Epidemiological and Economic Study quality of life and symptom (VEINES-QOL/Sym) questionnaires.
General health related quality of life | 3 months and 6 months
  General health related quality of life will be assessed by the 36-Item Short Form health questionnaire (SF-36).
  A high score corresponds to better health/quality of life.
Coagulation and fibrinolysis markers | up to 3 months
  D-dimers, plasminogen activator inhibitor 1 (PAI-1)
Fibrinolytic and pro-coagulant activities of microvesicles/microparticles | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ELIAS, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne-sur-Mer
Locations (23):
- France (23):
  - Centre Hospitalier de Carcassonne, Carcassonne, Aude
  - Hôpital d'Aubagne, Aubagne, Bouches-du-Rhône
  - Hôpital Saint Joseph, Marseille, Bouches-du-Rhône
  - Hôpital La Timone, AP-HM, Marseille, Bouches-du-Rhône
  - Cabinet libéral, Martigues, Bouches-du-Rhône
  - Cabinet libéral, Ajaccio, Corse-du-sud
  - CHU de Dijon, Dijon, Côte d'Or
  - CHU de Besançon, Besançon, Doubs
  - Centre Hospitalier Universitaire de Brest, Brest, Finistère
  - Clinique Rive Gauche, Toulouse, Haut-Garonne
  - Centre de Santé Polyvalent de UGESSAP, Montoir-de-Bretagne, Loire-Atlantique
  - CHU Saint Etienne, Saint-Priest-en-Jarez, Pays de la Loire Region
  - Hospices Civils de Lyon, Hôpital Edouard Herriot, Lyon, Rhône
  - Centre Hospitalier Universitaire Amiens Picardie, Amiens, Somme
  - Centre Hospitalier de Fréjus/Saint-Raphaël, Fréjus, Var
  - Polyclinique Les Fleurs, Ollioules, Var
  - Centre cardio-vasculaire Esterel, Saint-Raphaël, Var
  - Cabinet libéral, Sanary-sur-Mer, Var
  - Cabinet libéral, Six-Fours-les-Plages, Var
  - Centre Hospitalier Intercommunal Toulon La Seyne-sur-Mer, Toulon, Var
  - Centre Hospitalier d'Avignon, Avignon, Vaucluse
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Hôpital Saint Joseph, Paris

IPD SHARING:
Plan to Share IPD: No